CLINICAL TRIAL: NCT00038571
Title: Phase II Study of Proteasome Inhibitor PS-341 For Patients With Relapsed or Refractory B Cell Lymphomas Previously Treated With Chemotherapy
Brief Title: Proteasome Inhibitor PS-341 Relapsed or Refractory B Cell Lymphomas Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-596
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma, B-Cell
Keywords: Cancer; Relapsed; Refractory; B cell lymphoma; Proteasome Inhibitor; PS-341
MeSH Terms: conditions — Lymphoma, B-Cell; Neoplasms; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (mantle-cell lymphoma) (Experimental)
  Interventions: Drug: PS341 (Bortezomib)
- Arm B (other B-cell lymphomas) (Experimental)
  Interventions: Drug: PS341 (Bortezomib)

INTERVENTIONS:
Drug: PS341 (Bortezomib) — 1.5 mg/m2 intravenous (IV) bolus push over 3 to 5 seconds on days 1, 4, 8, and 11, followed by a 10-day rest for a 21-day cycle.
  Other Names: Velcade; LPD-341; MLN341; PS-341

SUMMARY:
Purpose of Phase II study for B-cell lymphoma using PS341: Evaluate efficacy and toxicity of bortezomib in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Patients were stratified, based on preclinical data, into arm A (mantle-cell lymphoma) or arm B (other B-cell lymphomas) without limitation in number of prior therapies. Bortezomib was administered as an intravenous push (1.5 mg/m2) on days 1, 4, 8, and 11 every 21 days for a maximum of six cycles.

ELIGIBILITY:
INCLUSION:

* Relapsed or Refractory B cell lymphoma.
* Zubrod status </= 3.
* Measurable disease.
* No anti-cancer treatment within past 3 weeks.
* ANC >= 1500/uL, Plt >/= 50,000, Bilirubin <2 mg/dL, SGPT <2.5xULN, creatinine <2. Patients with ANC>/1000, PLT>/30000 will be eligible if due to massive splenomegaly and/or BM involvement.
* HIV negative.
* No active CNS lymphoma.
* No serious intercurrent illness, active infections or cancer except basal cell carcinoma of the skin or in situ cervical carcinoma.
* Not eligible for treatment of a higher priority. Patients may be entered before BMT.
* No pregnancy & age bearing females must be practicing adequate contraception.
* Age > 16.

EXCLUSION:

* Patients with platelets <30x10(9)/L within 14 days before enrollment.
* Patients with ANC<1.0 x10(9)/L within 14 days before enrollment.
* Patients with peripheral neuropathy >/= grade 3 within 14 days before enrollment.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Response to PS-341 | Every two 21-day cycles
  Patient response evaluated according to criteria of Cheson et al. Endoscopy obtained every two cycles to evaluate response using Complete Response (CR), Partial Response (PR), Progressive Disease, or Stable Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fayad, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org